CLINICAL TRIAL: NCT01900990
Title: A Randomized Controlled Trial of Noninvasive Positive Pressure Ventilation for Weaning From Mechanical Ventilation in Tracheotomy Patients
Brief Title: Noninvasive Positive Pressure Ventilation for Difficult Weaning in Tracheotomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, resident physician, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQYKDXFSDYYY
Record Dates: First submitted 2010-07-26; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Respiratory Failure
Keywords: Noninvasive Positive Pressure Ventilation; Invasive Positive Pressure Ventilation; tracheotomy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noninvasive ventilation weaning (Experimental): Patients in this group were weaned by noninvasive ventilation
  Interventions: Device: Noninvasive ventilation weaning
- Conventional weaning (No Intervention): Patients in this group were weaned by conventional stratiges.

INTERVENTIONS:
Device: Noninvasive ventilation weaning — We adopt Noninvasive Positive Pressure Ventilation in tracheotomy patients by capping the tracheotomy tube and deflating the cuff
  Other Names: capping tracheotomy tube
  Arms: Noninvasive ventilation weaning

SUMMARY:
The investigators adopt Noninvasive Positive Pressure Ventilation for weaning in tracheotomy patients innovatively. The investigators randomly allocate the subjects into two groups. One group is weaned by traditional strategy. The other one is weaned by Noninvasive Positive Pressure Ventilation by plugging the tracheotomy tube and deflating the cuff.

DETAILED DESCRIPTION:
The investigators adopt Noninvasive Positive Pressure Ventilation for weaning in tracheotomy patients innovatively .If patients'conditions met our defined criterions, the investigators randomly allocate two groups. One group adopts traditional weaning strategy, the other adopts Noninvasive Positive Pressure Ventilation. If patients' condition deteriorated in group two, the investigators turned them to invasive positive pressure ventilation, until patients adapted in a satisfactory condition, the investigators shift them into Noninvasive Positive Pressure Ventilation. The investigators will extubate the tracheotomy tube, if patients are received Noninvasive Positive Pressure Ventilation more than 24 to 48 hours. After extubation, the investigators try to wean Noninvasive Positive Pressure Ventilation. Successful wean is defined weaning mechanical ventilation more than 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* tracheotomy mechanical ventilation patients

Exclusion Criteria:

* pregnancy
* respiratory and hemodynamic instability
* Recent oral，nasal，facial or cranial trauma or surgery
* contra-indications for nasal or facial mask (facial skin lesions,...)
* recent history of upper gastro-intestinal surgery
* recent history of myocardial infarction
* unconscious patients
* non cooperative patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Main end-point defined as total duration of mechanical ventilation | from admission to hospital to discharge from it or death
  The total duration of mechanical ventilation was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.

SECONDARY OUTCOMES:
duration of invasive mechanical ventilation | from admission to hospital to discharge from it or death
  The duration of invasive mechanical ventilation was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.
duration of extubation tracheotomy tube | from admission to hospital to discharge from it or death
  The duration of extubation tracheotomy tube was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.
total duration of mechanical ventilation (invasive and non invasive) | from admission to hospital to discharge from it or death
  The total duration of mechanical ventilation (invasive and non invasive) was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.
successful weaning rate | from admission to hospital to discharge from it or death
  The sucessful weaning rate was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.
ICU length of stay | from admission to hospital to discharge from it or death
  The ICU lentgh of stay was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.
hospital length of stay | from admission to hospital to discharge from it or death
  The hospital lentgh of stay was measured from the patient admitted to hospital to discharge from it or death, an expected average of 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Duan Jun, Principal Investigator — The First Affiliated Hospital,Chongqing Medical Univercity
Locations (1):
- The First Affiliated Hospital ,Chongqing Medical Univercity, Chongqing, Chongqing Municipality, China